CLINICAL TRIAL: NCT01493726
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ALKS 9072 in Subjects With Chronic Stable Schizophrenia
Brief Title: A Study of ALKS 9072 in Subjects With Chronic Stable Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK9072-002
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ALKS 9072, Low dose (Experimental)
  Interventions: Drug: ALKS 9072, Low dose
- ALKS 9072, Med dose (Experimental)
  Interventions: Drug: ALKS 9072, Med dose
- ALKS 9072, High dose (Experimental)
  Interventions: Drug: ALKS 9072, High dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 9072, Low dose — IM injection, given monthly
  Arms: ALKS 9072, Low dose
Drug: ALKS 9072, Med dose — IM injection, given monthly
  Arms: ALKS 9072, Med dose
Drug: ALKS 9072, High dose — IM injection, given monthly
  Arms: ALKS 9072, High dose
Drug: Placebo — Dosed matched placebo IM injection, given monthly
  Arms: Placebo

SUMMARY:
This study will determine the pharmacokinetics (PK), safety, and tolerability of ALKS 9072 (also known as ALKS 9070) after 4 monthly doses in adults with chronic stable schizophrenia.

DETAILED DESCRIPTION:
Three active treatment groups and a placebo group are planned. Randomization will be sequential by dose level across the sites with placebo assignments randomly inserted. Each subject's participation will be approximately 8 months, including screening, treatment period, and a 3-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic schizophrenia that is clinically stable
* Body mass index (BMI) between 18.5 and 35.0 kg/m2, inclusive
* Stable antipsychotic medication regimen for >/= 2 months before Screening
* Be willing and able to be confined to an inpatient clinical research unit for a total of 37 days during the course of the study

Exclusion Criteria:

* Aripiprazole used within 30 days before Screening
* History of intolerance of or allergy or hypersensitivity to aripiprazole, its excipients, other antipsychotic agents, or INTRALIPID (including peanuts, soy, egg, or glycerol)
* Current diagnosis of an Axis I disorder other than schizophrenia
* History of seizure disorder or any condition associated with seizures
* History of neuroleptic malignant syndrome (NMS)
* Positive test result for HIV, hepatitis B surface antigen, or anti-hepatitis C antibodies
* Received medication by IM injection within 30 days before Screening
* Monoamine oxidase inhibitors (eg, phenelzine, tranylcypromine, selegiline) used within 30 days before Screening
* DSM-IV-TR diagnosis of alcohol or substance dependence, with the exception of nicotine or caffeine dependence within 12 months before Screening
* Donation of blood or blood components within 4 weeks before Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration in plasma following last dose | 4 months
Time to maximum concentration in plasma following last dose | 4 months
Area under the plasma concentration time curve over the last dosing interval | 4 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, MD, Study Director — Alkermes, Inc.
Locations (6):
- United States (6):
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Willingboro, New Jersey
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Irving, Texas

REFERENCES:
- [Result] Hard ML, Mills RJ, Sadler BM, Turncliff RZ, Citrome L. Aripiprazole Lauroxil: Pharmacokinetic Profile of This Long-Acting Injectable Antipsychotic in Persons With Schizophrenia. J Clin Psychopharmacol. 2017 Jun;37(3):289-295. doi: 10.1097/JCP.0000000000000691. PMID 28350572